CLINICAL TRIAL: NCT05384535
Title: Utility of Biparametric MRI (Magnetic Resonance Imaging) as a Screening Tool for Prostate Cancer in a High-Risk Cohort
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwell Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 21-1380
Record Dates: First submitted 2022-05-17; First posted 2022-05-20 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Prostate Cancer; Magnetic Resonance Imaging; Population at Risk
Keywords: Prostate Cancer; Screening; Magnetic Resonance Imaging
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Bi-parametric Screening MRI (Experimental): Bi-parametric MRI to be administered to High Risk males
  Interventions: Diagnostic Test: Bi-parametric MRI

INTERVENTIONS:
Diagnostic Test: Bi-parametric MRI — When used for the evaluation of prostate cancer, MRI typically involves multiple sequences and typically includes typical T1 and T2 phases with the addition of diffusion weighted imaging and dynamic contrast enhanced imaging. In this study, we have decided to omit dynamic contrast enhanced imaging due to its decreased diagnostic yield relative to T2 and DWI and associated increased risk of contrast agents, this is a common approach for prostate cancer screening and is referred to as a bi-parametric MRI

SUMMARY:
To determine whether using bpMRI in subjects who are at high risk of developing prostate cancer in conjunction with PSA will improve prostate cancer screening protocols.

DETAILED DESCRIPTION:
The Investigators propose a pilot study which utilizes bpMRI in conjunction with PSA in the early detection of clinically significant prostate cancer in a high-risk group. Our study would focus on these high-risk subjects between the ages of 40-55 with a normal PSA ranging from ≥1.0 to <2.5 ng/mL. bpMRI would be obtained in this group of subjects. If any suspicious lesions are found, the recommendation is to undergo MRI/US fusion biopsy. Subjects with negative bpMRI will be followed every year with serum PSA. Subjects with a positive bpMRI will have a prostate fusion and systematic biopsy performed. Those with a benign biopsy will be followed every year with serum PSA. Those who have a biopsy positive for cancer will be managed and followed according to the standard of care. All subjects will be followed for 5 years. Our hypothesis is that bpMRI in conjunction with above average PSA in a high-risk group will increase detection of clinically relevant prostate cancer and provide a useful addition to PSA screening.

ELIGIBILITY:
Inclusion Criteria:

1. PSA between 1.0 and 2.5 ng/dL
2. High risk for prostate cancer, i.e. Black or they have a first degree relative with history of prostate cancer (father, brother) or specific genetic syndromes i.e. BRCA 1/2, HOX B13, Lynch syndrome, ATM, CHEK2
3. Patient is willing to participated in prostate cancer screening
4. Patient is capable of giving informed consent

Exclusion Criteria:

1. Nodularity or firmness of prostate on exam
2. Patient has undergone a prior biopsy or prostate surgery
3. Patient is taking 5-alpha reductase inhibitors to manage benign prostatic hyperplasia, as this can significantly alter PSA levels.
4. Patient has a history of UTI or prostatitis in the preceding 6 months, as this can significantly alter PSA levels.
5. Patient has a contraindication to MRI, these include but are not limited to pacemakers, neurostimulator devices, metal cardiac valves, certain tattoos, or foreign bodies
6. Participants that experience claustrophobia, anxiety and/or vertigo when moved inside the scanner
7. The participant cannot tolerate lying flat for the study duration

Ages: 40 Years to 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-08-15 (Actual); Primary Completion 2027-10-31 (Estimated); Study Completion 2028-10-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of suspicious lesions on MRI in men with PSA less than 2.5 ng/ml | 3 months
  To determine the incidence of positive mpMRI prostate in a high-risk cohort of men as a screening tool for prostate cancer.

SECONDARY OUTCOMES:
Prostate cancer detection rate using 3T bpMRI in patients with high risk and suspicious lesions on bpMRI | 3 months
  Proportion of men with suspicious lesion found to have cancer on biopsy, this is the PPV based on the prevalence of this population.
Association of whether findings on bpMRI and serum PSA (i.e. PSA density) are associated with future diagnosis of prostate cancer. | 5 years
  Proportion diagnosed with prostate cancer over 5 year follow-up among patients who were not diagnosed with prostate cancer based on findings of initial mpMRI (i.e. mend who either did not have any suspicious lesions or had suspicious lesions but were negative for cancer on biopsy)
To correlate bpMRI findings with future changes in PSA | 5 years
  PSA density will be measured every year for five years

CONTACTS AND LOCATIONS:
Overall Officials: Ardeshir Rastinehad, DO, Principal Investigator — Northwell Health; Manish Vira, MD, Principal Investigator — Northwell Health
Locations (1):
- Cynthia Knauer, Lake Success, New York, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD with other researchers

REFERENCES:
- [Background] Sanda MG, Cadeddu JA, Kirkby E, Chen RC, Crispino T, Fontanarosa J, Freedland SJ, Greene K, Klotz LH, Makarov DV, Nelson JB, Rodrigues G, Sandler HM, Taplin ME, Treadwell JR. Clinically Localized Prostate Cancer: AUA/ASTRO/SUO Guideline. Part I: Risk Stratification, Shared Decision Making, and Care Options. J Urol. 2018 Mar;199(3):683-690. doi: 10.1016/j.juro.2017.11.095. Epub 2017 Dec 15. PMID 29203269
- [Background] Qaseem A, Barry MJ, Denberg TD, Owens DK, Shekelle P; Clinical Guidelines Committee of the American College of Physicians. Screening for prostate cancer: a guidance statement from the Clinical Guidelines Committee of the American College of Physicians. Ann Intern Med. 2013 May 21;158(10):761-769. doi: 10.7326/0003-4819-158-10-201305210-00633. PMID 23567643
- [Background] Mohler JL, Antonarakis ES, Armstrong AJ, D'Amico AV, Davis BJ, Dorff T, Eastham JA, Enke CA, Farrington TA, Higano CS, Horwitz EM, Hurwitz M, Ippolito JE, Kane CJ, Kuettel MR, Lang JM, McKenney J, Netto G, Penson DF, Plimack ER, Pow-Sang JM, Pugh TJ, Richey S, Roach M, Rosenfeld S, Schaeffer E, Shabsigh A, Small EJ, Spratt DE, Srinivas S, Tward J, Shead DA, Freedman-Cass DA. Prostate Cancer, Version 2.2019, NCCN Clinical Practice Guidelines in Oncology. J Natl Compr Canc Netw. 2019 May 1;17(5):479-505. doi: 10.6004/jnccn.2019.0023. PMID 31085757
- [Background] Catalona WJ, Smith DS, Ratliff TL, Dodds KM, Coplen DE, Yuan JJ, Petros JA, Andriole GL. Measurement of prostate-specific antigen in serum as a screening test for prostate cancer. N Engl J Med. 1991 Apr 25;324(17):1156-61. doi: 10.1056/NEJM199104253241702. PMID 1707140
- [Background] Hofbauer SL, Maxeiner A, Kittner B, Heckmann R, Reimann M, Wiemer L, Asbach P, Haas M, Penzkofer T, Stephan C, Friedersdorff F, Fuller F, Miller K, Cash H. Validation of Prostate Imaging Reporting and Data System Version 2 for the Detection of Prostate Cancer. J Urol. 2018 Oct;200(4):767-773. doi: 10.1016/j.juro.2018.05.003. Epub 2018 May 5. PMID 29733838
- [Background] Ahmed HU, El-Shater Bosaily A, Brown LC, Gabe R, Kaplan R, Parmar MK, Collaco-Moraes Y, Ward K, Hindley RG, Freeman A, Kirkham AP, Oldroyd R, Parker C, Emberton M; PROMIS study group. Diagnostic accuracy of multi-parametric MRI and TRUS biopsy in prostate cancer (PROMIS): a paired validating confirmatory study. Lancet. 2017 Feb 25;389(10071):815-822. doi: 10.1016/S0140-6736(16)32401-1. Epub 2017 Jan 20. PMID 28110982
- [Background] Siegel R, Naishadham D, Jemal A. Cancer statistics, 2012. CA Cancer J Clin. 2012 Jan-Feb;62(1):10-29. doi: 10.3322/caac.20138. Epub 2012 Jan 4. PMID 22237781
- [Background] Zhen JT, Syed J, Nguyen KA, Leapman MS, Agarwal N, Brierley K, Llor X, Hofstatter E, Shuch B. Genetic testing for hereditary prostate cancer: Current status and limitations. Cancer. 2018 Aug 1;124(15):3105-3117. doi: 10.1002/cncr.31316. Epub 2018 Apr 18. PMID 29669169
- [Background] Vickers AJ, Ulmert D, Sjoberg DD, Bennette CJ, Bjork T, Gerdtsson A, Manjer J, Nilsson PM, Dahlin A, Bjartell A, Scardino PT, Lilja H. Strategy for detection of prostate cancer based on relation between prostate specific antigen at age 40-55 and long term risk of metastasis: case-control study. BMJ. 2013 Apr 15;346:f2023. doi: 10.1136/bmj.f2023. PMID 23596126
- [Background] Hu Y, Ahmed HU, Carter T, Arumainayagam N, Lecornet E, Barzell W, Freeman A, Nevoux P, Hawkes DJ, Villers A, Emberton M, Barratt DC. A biopsy simulation study to assess the accuracy of several transrectal ultrasonography (TRUS)-biopsy strategies compared with template prostate mapping biopsies in patients who have undergone radical prostatectomy. BJU Int. 2012 Sep;110(6):812-20. doi: 10.1111/j.1464-410X.2012.10933.x. Epub 2012 Mar 6. PMID 22394583
- [Background] Fleshner NE, O'Sullivan M, Fair WR. Prevalence and predictors of a positive repeat transrectal ultrasound guided needle biopsy of the prostate. J Urol. 1997 Aug;158(2):505-8; discussion 508-9. PMID 9224334
- [Background] Brown LC, Ahmed HU, Faria R, El-Shater Bosaily A, Gabe R, Kaplan RS, Parmar M, Collaco-Moraes Y, Ward K, Hindley RG, Freeman A, Kirkham A, Oldroyd R, Parker C, Bott S, Burns-Cox N, Dudderidge T, Ghei M, Henderson A, Persad R, Rosario DJ, Shergill I, Winkler M, Soares M, Spackman E, Sculpher M, Emberton M. Multiparametric MRI to improve detection of prostate cancer compared with transrectal ultrasound-guided prostate biopsy alone: the PROMIS study. Health Technol Assess. 2018 Jul;22(39):1-176. doi: 10.3310/hta22390. PMID 30040065
- [Background] Drost FH, Osses DF, Nieboer D, Steyerberg EW, Bangma CH, Roobol MJ, Schoots IG. Prostate MRI, with or without MRI-targeted biopsy, and systematic biopsy for detecting prostate cancer. Cochrane Database Syst Rev. 2019 Apr 25;4(4):CD012663. doi: 10.1002/14651858.CD012663.pub2. PMID 31022301
- [Background] Elwenspoek MMC, Sheppard AL, McInnes MDF, Merriel SWD, Rowe EWJ, Bryant RJ, Donovan JL, Whiting P. Comparison of Multiparametric Magnetic Resonance Imaging and Targeted Biopsy With Systematic Biopsy Alone for the Diagnosis of Prostate Cancer: A Systematic Review and Meta-analysis. JAMA Netw Open. 2019 Aug 2;2(8):e198427. doi: 10.1001/jamanetworkopen.2019.8427. PMID 31390032
- [Background] Weinrich SP. Prostate cancer screening in high-risk men: African American Hereditary Prostate Cancer Study Network. Cancer. 2006 Feb 15;106(4):796-803. doi: 10.1002/cncr.21674. PMID 16411222
- [Background] Martin AJ, Lord SJ, Verry HE, Stockler MR, Emery JD. Risk assessment to guide prostate cancer screening decisions: a cost-effectiveness analysis. Med J Aust. 2013 Jun 3;198(10):546-50. doi: 10.5694/mja12.11597. PMID 23725269
- [Background] Leach MO, Brindle KM, Evelhoch JL, Griffiths JR, Horsman MR, Jackson A, Jayson GC, Judson IR, Knopp MV, Maxwell RJ, McIntyre D, Padhani AR, Price P, Rathbone R, Rustin GJ, Tofts PS, Tozer GM, Vennart W, Waterton JC, Williams SR, Workman P; Pharmacodynamic/Pharmacokinetic Technologies Advisory Committee, Drug Development Office, Cancer Research UK. The assessment of antiangiogenic and antivascular therapies in early-stage clinical trials using magnetic resonance imaging: issues and recommendations. Br J Cancer. 2005 May 9;92(9):1599-610. doi: 10.1038/sj.bjc.6602550. PMID 15870830
- [Background] Padhani AR, Liu G, Koh DM, Chenevert TL, Thoeny HC, Takahara T, Dzik-Jurasz A, Ross BD, Van Cauteren M, Collins D, Hammoud DA, Rustin GJ, Taouli B, Choyke PL. Diffusion-weighted magnetic resonance imaging as a cancer biomarker: consensus and recommendations. Neoplasia. 2009 Feb;11(2):102-25. doi: 10.1593/neo.81328. PMID 19186405
- [Background] Le Bihan D, Turner R, Douek P, Patronas N. Diffusion MR imaging: clinical applications. AJR Am J Roentgenol. 1992 Sep;159(3):591-9. doi: 10.2214/ajr.159.3.1503032.
- [Background] Le Bihan D, Douek P, Argyropoulou M, Turner R, Patronas N, Fulham M. Diffusion and perfusion magnetic resonance imaging in brain tumors. Top Magn Reson Imaging. 1993 Winter;5(1):25-31. PMID 8416686
- [Background] Koh DM, Collins DJ. Diffusion-weighted MRI in the body: applications and challenges in oncology. AJR Am J Roentgenol. 2007 Jun;188(6):1622-35. doi: 10.2214/AJR.06.1403. PMID 17515386
- [Background] Chandarana H, Taouli B. Diffusion-weighted MRI and liver metastases. Magn Reson Imaging Clin N Am. 2010 Aug;18(3):451-64, x. doi: 10.1016/j.mric.2010.07.001. PMID 21094449
- [Background] Nasu K, Kuroki Y, Tsukamoto T, Nakajima H, Mori K, Minami M. Diffusion-weighted imaging of surgically resected hepatocellular carcinoma: imaging characteristics and relationship among signal intensity, apparent diffusion coefficient, and histopathologic grade. AJR Am J Roentgenol. 2009 Aug;193(2):438-44. doi: 10.2214/AJR.08.1424. PMID 19620441
- [Background] Belli P, Costantini M, Bufi E, Magistrelli A, La Torre G, Bonomo L. Diffusion-weighted imaging in breast lesion evaluation. Radiol Med. 2010 Feb;115(1):51-69. doi: 10.1007/s11547-009-0430-6. Epub 2009 Nov 9. English, Italian. PMID 19902330
- [Background] Hoeks CM, Barentsz JO, Hambrock T, Yakar D, Somford DM, Heijmink SW, Scheenen TW, Vos PC, Huisman H, van Oort IM, Witjes JA, Heerschap A, Futterer JJ. Prostate cancer: multiparametric MR imaging for detection, localization, and staging. Radiology. 2011 Oct;261(1):46-66. doi: 10.1148/radiol.11091822. PMID 21931141
- [Background] Hankey BF, Feuer EJ, Clegg LX, Hayes RB, Legler JM, Prorok PC, Ries LA, Merrill RM, Kaplan RS. Cancer surveillance series: interpreting trends in prostate cancer--part I: Evidence of the effects of screening in recent prostate cancer incidence, mortality, and survival rates. J Natl Cancer Inst. 1999 Jun 16;91(12):1017-24. doi: 10.1093/jnci/91.12.1017. PMID 10379964
- [Background] Baquet CR, Horm JW, Gibbs T, Greenwald P. Socioeconomic factors and cancer incidence among blacks and whites. J Natl Cancer Inst. 1991 Apr 17;83(8):551-7. doi: 10.1093/jnci/83.8.551. PMID 2005640
- [Background] Platz EA, Rimm EB, Willett WC, Kantoff PW, Giovannucci E. Racial variation in prostate cancer incidence and in hormonal system markers among male health professionals. J Natl Cancer Inst. 2000 Dec 20;92(24):2009-17. doi: 10.1093/jnci/92.24.2009. PMID 11121463
- [Background] Odedina FT, Akinremi TO, Chinegwundoh F, Roberts R, Yu D, Reams RR, Freedman ML, Rivers B, Green BL, Kumar N. Prostate cancer disparities in Black men of African descent: a comparative literature review of prostate cancer burden among Black men in the United States, Caribbean, United Kingdom, and West Africa. Infect Agent Cancer. 2009 Feb 10;4 Suppl 1(Suppl 1):S2. doi: 10.1186/1750-9378-4-S1-S2. PMID 19208207
- [Background] Parker PM, Rice KR, Sterbis JR, Chen Y, Cullen J, McLeod DG, Brassell SA. Prostate cancer in men less than the age of 50: a comparison of race and outcomes. Urology. 2011 Jul;78(1):110-5. doi: 10.1016/j.urology.2010.12.046. Epub 2011 Mar 12. PMID 21397300
- [Background] Hoffman RM, Gilliland FD, Eley JW, Harlan LC, Stephenson RA, Stanford JL, Albertson PC, Hamilton AS, Hunt WC, Potosky AL. Racial and ethnic differences in advanced-stage prostate cancer: the Prostate Cancer Outcomes Study. J Natl Cancer Inst. 2001 Mar 7;93(5):388-95. doi: 10.1093/jnci/93.5.388. PMID 11238701
- [Background] Mahal BA, Aizer AA, Ziehr DR, Hyatt AS, Sammon JD, Schmid M, Choueiri TK, Hu JC, Sweeney CJ, Beard CJ, D'Amico AV, Martin NE, Kim SP, Trinh QD, Nguyen PL. Trends in disparate treatment of African American men with localized prostate cancer across National Comprehensive Cancer Network risk groups. Urology. 2014 Aug;84(2):386-92. doi: 10.1016/j.urology.2014.05.009. Epub 2014 Jun 26. PMID 24975710
- [Background] Barocas DA, Penson DF. Racial variation in the pattern and quality of care for prostate cancer in the USA: mind the gap. BJU Int. 2010 Aug;106(3):322-8. doi: 10.1111/j.1464-410X.2010.09467.x. Epub 2010 Jun 14. PMID 20553251
- [Background] Bratt O, Drevin L, Akre O, Garmo H, Stattin P. Family History and Probability of Prostate Cancer, Differentiated by Risk Category: A Nationwide Population-Based Study. J Natl Cancer Inst. 2016 Jul 10;108(10):djw110. doi: 10.1093/jnci/djw110. Print 2016 Oct. PMID 27400876
- [Background] Madersbacher S, Alcaraz A, Emberton M, Hammerer P, Ponholzer A, Schroder FH, Tubaro A. The influence of family history on prostate cancer risk: implications for clinical management. BJU Int. 2011 Mar;107(5):716-721. doi: 10.1111/j.1464-410X.2010.10024.x. Epub 2010 Dec 16. PMID 21166744
- [Background] Jambor I, Verho J, Ettala O, Knaapila J, Taimen P, Syvanen KT, Kiviniemi A, Kahkonen E, Perez IM, Seppanen M, Rannikko A, Oksanen O, Riikonen J, Vimpeli SM, Kauko T, Merisaari H, Kallajoki M, Mirtti T, Lamminen T, Saunavaara J, Aronen HJ, Bostrom PJ. Validation of IMPROD biparametric MRI in men with clinically suspected prostate cancer: A prospective multi-institutional trial. PLoS Med. 2019 Jun 3;16(6):e1002813. doi: 10.1371/journal.pmed.1002813. eCollection 2019 Jun. PMID 31158230
- [Background] Bass EJ, Pantovic A, Connor M, Gabe R, Padhani AR, Rockall A, Sokhi H, Tam H, Winkler M, Ahmed HU. A systematic review and meta-analysis of the diagnostic accuracy of biparametric prostate MRI for prostate cancer in men at risk. Prostate Cancer Prostatic Dis. 2021 Sep;24(3):596-611. doi: 10.1038/s41391-020-00298-w. Epub 2020 Nov 20. PMID 33219368
- [Background] Qiao EM, Lynch JA, Lee KM, Kotha NV, Nalawade V, Voora RS, Qian AS, Nelson TJ, Yamoah K, Garraway IP, Stewart TF, Parsons JK, Rose BS. Evaluating Prostate-Specific Antigen Screening for Young African American Men With Cancer. J Natl Cancer Inst. 2022 Apr 11;114(4):592-599. doi: 10.1093/jnci/djab221. PMID 34893859
- See also: Guidance for Industry and FDA Staff: Criteria for Significant Risk Investigations of Magnetic Resonance Diagnostic Devices — https://www.fda.gov/media/71385/download
- See also: Medical Device Regulation and Overview General and Special Controls — http://www.fda.gov/MedicalDevices/DeviceRegulationandGuidance/Overview/GeneralandSpecialControls/ucm055910.htm
- See also: How to Market Your Device — http://www.fda.gov/MedicalDevices/DeviceRegulationandGuidance/HowtoMarketYourDevice/RegistrationandListing/ucm053165.htm
- See also: How to market Your Device (2) — http://www.fda.gov/MedicalDevices/DeviceRegulationandGuidance/HowtoMarketYourDevice/RegistrationandListing/ucm053156.htm
- See also: Accessing Data — http://www.accessdata.fda.gov/scripts/cdrh/cfdocs/cfRL/rl.cfm
- See also: Post Market Regulation Requirements — http://www.fda.gov/MedicalDevices/DeviceRegulationandGuidance/PostmarketRequirements/QualitySystemsRegulations/default.htm